CLINICAL TRIAL: NCT06952803
Title: A Randomised, Double-blind, Placebo-controlled, Phase III Study of Adjuvant Saruparib (AZD5305) in Patients With BRCAm Localised High-Risk Prostate Cancer Receiving Radiotherapy With Androgen Deprivation Therapy (EvoPAR-Prostate02).
Brief Title: A Study of Metastases Free Survival With Saruparib vs Placebo Added to a Standard RT/ADT in Men With High-risk Prostate Cancer With a BRCA Mutation
Acronym: EvoPAR-PR02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9727C00001; 2024-513586-39 (Other: EU CT Number)
Record Dates: First submitted 2025-04-30; First posted 2025-05-01 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: Localised/locally advanced prostate cancer; High-risk biochemical recurrence (BCR); Poly (ADP-ribose) polymerase; Radiation therapy or radiotherapy; Breast cancer gene (BRCA) mutation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — AZD5305; abiraterone; Prednisolone; Prednisone; Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: Saruparib (AZD5305) + Physician's Choice ADT (Experimental): Participants will receive saruparib along with ADT.
  Interventions: Drug: Saruparib; Drug: Androgen Deprivation Therapy (ADT)
- Cohort A: Placebo + Physician's Choice ADT (Placebo Comparator): Participants will receive matching placebo to saruparib along with ADT.
  Interventions: Drug: Placebo; Drug: Androgen Deprivation Therapy (ADT)
- Cohort B: Saruparib (AZD5305) + Physician's Choice ADT + Abiraterone (and prednisone/prednisolone) (Experimental): Participants will receive saruparib, abiraterone and prednisolone/prednisone along with ADT.
  Interventions: Drug: Saruparib; Drug: Abiraterone + Prednisolone/Prednisone; Drug: Androgen Deprivation Therapy (ADT)
- Cohort B: Placebo + Physician's Choice ADT + Abiraterone (and prednisone/prednisolone) (Placebo Comparator): Participants will receive matching placebo to saruparib, abiraterone and prednisolone/prednisone along with ADT.
  Interventions: Drug: Placebo; Drug: Abiraterone + Prednisolone/Prednisone; Drug: Androgen Deprivation Therapy (ADT)

INTERVENTIONS:
Drug: Saruparib — Saruparib will be administered orally.
  Other Names: AZD5305
  Arms: Cohort A: Saruparib (AZD5305) + Physician's Choice ADT; Cohort B: Saruparib (AZD5305) + Physician's Choice ADT + Abiraterone (and prednisone/prednisolone)
Drug: Placebo — Matching placebo to saruparib will be administered orally.
  Arms: Cohort A: Placebo + Physician's Choice ADT; Cohort B: Placebo + Physician's Choice ADT + Abiraterone (and prednisone/prednisolone)
Drug: Abiraterone + Prednisolone/Prednisone — Abiraterone will be administered orally in combination with prednisone/prednisolone.
  Arms: Cohort B: Placebo + Physician's Choice ADT + Abiraterone (and prednisone/prednisolone); Cohort B: Saruparib (AZD5305) + Physician's Choice ADT + Abiraterone (and prednisone/prednisolone)
Drug: Androgen Deprivation Therapy (ADT) — Standard of care ADT will be administered.

SUMMARY:
The purpose of the study is to demonstrate superiority of Saruparib (AZD5305) relative to placebo added to a standard radiation therapy (RT) + androgen deprivation therapy (ADT) regimen by assessment of metastases-free survival in participants with high-risk and very high-risk localised/locally advanced prostate cancer with a breast cancer gene mutation (BRCAm).

DETAILED DESCRIPTION:
Approximately, 700 adult participants with localised/locally advanced prostate cancer will be randomized in a 1:1 ratio to receive saruparib or placebo with ADT (+ abiraterone) in one of the following two cohorts:

Cohort A: 400 adult participants with newly diagnosed high-risk and very high-risk (localised/locally advanced) prostate cancer who have received primary RT and are receiving continuous ADT, and participants with high-risk biochemical recurrence (BCR) [including prostate-specific antigen (PSA) persistence] following a radical prostatectomy who have received salvage RT are receiving continuous ADT.

Cohort B: 300 adult participants with newly diagnosed very high-risk (locally advanced) prostate cancer who have received primary RT and who are receiving continuous ADT and abiraterone.

All participants will be followed for survival until the end of the study. Independent data monitoring committee (DMC) composed of experts will be convened to confirm the safety and efficacy of Saruparib + ADT (+ abiraterone).

ELIGIBILITY:
Inclusion Criteria:

* Male participants with a histologically documented diagnosis of prostate adenocarcinoma.
* Newly diagnosed high-risk and very high-risk (localised/locally advanced) prostate cancer or a high-risk biochemical recurrence (BCR) following radical prostatectomy.
* Provision of a formalin fixed and paraffin embedded (FFPE) tumour tissue sample.
* Confirmed BRCA1 or BRCA2 mutation status by central tumour tissue is required for enrolment.
* Participants required to have a computed tomography (CT) or magnetic resonance imaging (MRI) and a bone scan following the completion of their planned RT. This screening scan must confirm no evidence of disease or evidence of disease confined to the pelvis (M0).
* Participants required to have a prostate-specific membrane antigen-positron emission tomography (PSMA-PET) following the completion of their planned RT. This screening scan must confirm no evidence of disease or evidence of disease confined to the pelvis (M0).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration over the 2 weeks prior to randomization.
* Minimum life expectancy of 12 months.
* Adequate organ and bone marrow function as described in study protocol.
* All participants will have received either primary or salvage RT. Participants must be eligible for randomisation within 10 months of initial diagnosis (de novo or BCR). Radiotherapy administered to the prostate (± pelvis) either in the primary or salvage setting must be delivered with curative intent. Use of metastases-directed therapy, as part of the RT radiation plan, is permitted as localised RT treatment for a metastatic lesion(s) outside the pelvis.
* All participants will have received a planned regimen of ADT with a gonadotropin releasing hormone (GnRH) analogue.
* Participants must not father children or donate sperm from signing informed consent form (ICF), during the study intervention and for 6 months after the last dose of study intervention.
* Participants must use a condom (with spermicide - where permitted) from signing ICF, during study intervention, and for 6 months after the last dose of study drug, with all sexual partners.

Exclusion Criteria:

* Participants with a history of myelodysplastic syndrome (MDS)/ acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* Participants with any known predisposition to bleeding [e.g., active peptic ulceration, recent (within 6 months) hemorrhagic stroke, proliferative diabetic retinopathy].
* Any history of persisting (> 2 weeks) severe cytopenia due to any cause.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of saruparib and/or abiraterone.
* History of another primary malignancy, with exceptions.
* Persistent toxicities [Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥ 2] caused by previous anticancer therapy.
* Cardiac criteria, including history of arrhythmia and cardiovascular disease.
* Evidence of active and uncontrolled hepatitis B and/or hepatitis C.
* Evidence of active and uncontrolled human immunodeficiency virus (HIV) infection.
* Active tuberculosis infection.
* Any prior chemotherapy (i.e., docetaxel) or immunotherapy; any prior treatment with a poly (ADP-ribose) polymerase (PARP) inhibitor.
* Prior treatment within 14 days with blood product support or growth factor support.
* Concomitant use of strong inducers and inhibitors of CYP3A4 (applies to saruparib and abiraterone) or herbal supplements within 21 days or at least 5 half-lives (whichever is longer), of randomization.
* Concomitant use of drugs that are known to prolong QT and have a known risk of Torsades de Pointes (TdP).
* Participants with a known hypersensitivity to saruparib or any excipients of these products.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 700 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2033-03-31 (Estimated); Study Completion 2036-04-30 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival (MFS) | Up to approximately 93 months
  MFS is defined as the time from randomisation until the date of first appearance of distant metastases, confirmed by standard clinical imaging [computed tomography (CT)/ magnetic resonance imaging (MRI) and bone scan, or prostate-specific membrane antigen-positron emission tomography (PSMA-PET)], as assessed by blinded independent central review (BICR) or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 11 years
  OS is defined as the time from randomisation until the date of death due to any cause.
MFS (CT/MRI and bone scan) | Up to approximately 93 months
  MFS is defined as the time from randomisation until the date of distant metastases, confirmed by conventional imaging (CT/MRI and bone scan), or death due to any cause.
MFS (PSMA-PET) | Up to approximately 93 months
  MFS is defined as the time from randomisation until the date of distant metastases, confirmed by PSMA-PET imaging or death due to any cause.
MFS (standard clinical imaging) | Up to approximately 93 months
  MFS is defined as the time from randomisation until the date of distant metastases, confirmed by standard clinical imaging (CT/MRI and bone scan or PSMA-PET), histology, or death due to any cause.
Time from randomisation to Progression Free Survival 2 (PFS2) | Up to approximately 93 months
  Time from randomisation to PFS2 is defined as the time from randomisation to the earliest of progression [defined as radiographic progression, clinical progression, or prostate-specific antigen (PSA) progression] after initiation of first subsequent systemic treatment following the initial investigator-assessed progression or death. The date of second progression will be investigator assessed according to local standard clinical practice.
Time to biochemical recurrence | Up to approximately 93 months
  Time to biochemical recurrence is defined as the time from randomisation to biochemical recurrence per Phoenix criteria.
Prostate cancer-specific survival (PCSS) | Up to approximately 11 years
  PCSS is defined as the time from randomisation until the date of death due to the underlying prostate cancer.
Time to deterioration in urinary symptoms (TTDUS) | Up to approximately 93 months
  TTDUS is defined as the time from randomisation to deterioration in EORTC-QLQ-PR25 (US) subscale scores.
Time to deterioration in physical function (TTDPF) | Up to approximately 93 months
  TTDPF is defined as the time from randomisation to deterioration in EORTC-QLQ-C30 Physical Function subscale scores.
Plasma concentrations of saruparib | Day 1 of Cycle 1, Cycle 3 and Cycle 6 (each cycle is of 28 days)
  To assess the PK of saruparib in plasma either with or without abiraterone and explore the relationship between the PK concentration/parameters and selected endpoints (which may include pharmacodynamic parameters, efficacy, and/or safety).
Area under the curve (AUC) | Day 1 of Cycle 1, Cycle 3 and Cycle 6 (each cycle is of 28 days)
  To assess the PK of saruparib in plasma either with or without abiraterone and explore the relationship between the PK concentration/parameters and selected endpoints (which may include pharmacodynamic parameters, efficacy, and/or safety).
Maximum observed concentration (Cmax) | Day 1 of Cycle 1, Cycle 3 and Cycle 6 (each cycle is of 28 days)
  To assess the PK of saruparib in plasma either with or without abiraterone and explore the relationship between the PK concentration/parameters and selected endpoints (which may include pharmacodynamic parameters, efficacy, and/or safety).
Time to Cmax (Tmax) | Day 1 of Cycle 1, Cycle 3 and Cycle 6 (each cycle is of 28 days)
  To assess the PK of saruparib in plasma either with or without abiraterone and explore the relationship between the PK concentration/parameters and selected endpoints (which may include pharmacodynamic parameters, efficacy, and/or safety).
Number of participants with adverse events (AEs) | Up to approximately 11 years
  To assess the safety and tolerability of saruparib administered in combination with ADT alone (Cohort A) and in combination with ADT + abiraterone (Cohort B).

CONTACTS AND LOCATIONS:
Locations (267):
- United States (39):
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, San Luis Obispo, California
  - Research Site, Lakewood, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Newnan, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Chicago Ridge, Illinois
  - Research Site, Greenwood, Indiana
  - Research Site, Jeffersonville, Indiana
  - Research Site, Bethesda, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Plymouth, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Hackensack, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, New York, New York
  - Research Site, Syracuse, New York
  - Research Site, Columbus, Ohio
  - Research Site, Springfield, Oregon
  - Research Site, Hershey, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Spring, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Seattle, Washington
- Argentina (8):
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Cuidad Autónoma de Buenos Aire
  - Research Site, La Plata
  - Research Site, Pergamino
  - Research Site, San Miguel de Tucumán
  - Research Site, Viedma
- Australia (7):
  - Research Site, Kingswood
  - Research Site, Murdoch
  - Research Site, Orange
  - Research Site, South Brisbane
  - Research Site, St Leonards
  - Research Site, Waratah
  - Research Site, Woolloongabba
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (6):
  - Research Site, Brussels
  - Research Site, Jette
  - Research Site, Kortrijk
  - Research Site, Libramont-Chevigny
  - Research Site, Roeselare
  - Research Site, Wilrijk
- Brazil (9):
  - Research Site, Cachoeiro de Itapemirim
  - Research Site, Curitiba
  - Research Site, Jaú
  - Research Site, Londrina
  - Research Site, Pelotas
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Abbotsford, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Barrie, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, London, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Toronto
- Chile (2):
  - Research Site, Concepción
  - Research Site, Temuco
- China (20):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Sichuan
  - Research Site, Suining
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Wuhu
  - Research Site, Xiamen
  - Research Site, Yangzhou
  - Research Site, Zhuhai
- Finland (5):
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Oulu
  - Research Site, Tampere
  - Research Site, Turku
- France (19):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Le Mans
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
  - Research Site, Saint-Herblain
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Tours
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Germany (23):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Braunschweig
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Giessen
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, Herne
  - Research Site, Kiel
  - Research Site, Lübeck
  - Research Site, Marburg
  - Research Site, Münster
  - Research Site, Nuremberg
  - Research Site, Nürtingen
  - Research Site, Regensburg
  - Research Site, Schwerin
  - Research Site, Trier
  - Research Site, Ulm
  - Research Site, Würzburg
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Zalaegerszeg
- India (8):
  - Research Site, Ansārinagar
  - Research Site, Babgalore
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Kannur
  - Research Site, Mumbai
  - Research Site, Nagpur
  - Research Site, Varanasi
- Israel (8):
  - Research Site, Afula
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (14):
  - Research Site, Arezzo
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Chieti
  - Research Site, Genoa
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Torino
  - Research Site, Varese
  - Research Site, Verona
- Japan (13):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Kamakura-shi
  - Research Site, Kawagoe-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kisarazu-shi
  - Research Site, Kumamoto
  - Research Site, Maebashi
  - Research Site, Miyazaki
  - Research Site, Ōta-ku
  - Research Site, Sagamihara-shi
  - Research Site, Shimotsuke-shi
  - Research Site, Yokohama
- Malaysia (4):
  - Research Site, Batu Caves
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Pulau Pinang
- Netherlands (5):
  - Research Site, Hilversum
  - Research Site, Hoofddorp
  - Research Site, Maastricht
  - Research Site, Nijmegen
  - Research Site, Roosendaal
- Peru (2):
  - Research Site, Lima
  - Research Site, Trujillo
- Poland (8):
  - Research Site, Gdynia
  - Research Site, Gliwice
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Piotrkow Trybunalski
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Warsaw
- South Korea (4):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Sabadell
  - Research Site, Santander
  - Research Site, Valencia
- Sweden (5):
  - Research Site, Gothenburg
  - Research Site, Malmo
  - Research Site, Stockholm
  - Research Site, Umeå
  - Research Site, Uppsala
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Khon Kaen
  - Research Site, Muang
  - Research Site, Pathum Thani
  - Research Site, Songkhla
- Turkey (Türkiye) (7):
  - Research Site, Ankara
  - Research Site, Diyarbakır
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Karşıyaka
  - Research Site, Sakarya
  - Research Site, Şahinbey
- United Kingdom (15):
  - Research Site, Aberdeen
  - Research Site, Barnet
  - Research Site, Bristol
  - Research Site, Cambridge
  - Research Site, Edinburgh
  - Research Site, Exeter
  - Research Site, Glasgow
  - Research Site, Greater London
  - Research Site, Guildford
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle
  - Research Site, Plymouth
  - Research Site, Preston
  - Research Site, Romford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/